CLINICAL TRIAL: NCT05841420
Title: A Randomized Phase II Study of Gemcitabine Versus Reduced-dose Combination Chemotherapy in Fragile Patients with Non-resectable Pancreatic Cancer
Brief Title: Gemcitabine Versus Reduced-dose Combination Chemotherapy in Fragile Patients with Non-resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Morten Ladekarl (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Herlev and Gentofte Hospital (Other); Gødstrup Hospital (Other); Vejle Hospital (Other)
Responsible Party: Sponsor-Investigator, Morten Ladekarl, Professor, MD, Phd, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPCG-01
Record Dates: First submitted 2023-03-16; First posted 2023-05-03 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Pancreas Cancer; Non-Resectable Pancreas Carcinoma
Keywords: Fragile; Elderly; Palliative
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: "Full dose single agent strategy" (Active Comparator): Gemcitabine monotherapy, 1000 mg/m2 weekly on days 1, 8, and 15 every 4 weeks
  Interventions: Drug: Gemcitabine
- B: "Reduced dose (80%) combination-therapy strategy" (Experimental): Nab-Paclitaxel: 100mg/m2 plus gemcitabine: 800 mg/m2 on day 1, 8 and 15 every 4 weeks
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine monotherapy, 1000 mg/m2 weekly on days 1, 8, and 15 every 4 weeks or gemcitabine: 800 mg/m2 on day 1, 8 and 15 every 4 weeks
  Other Names: Gemzar
Drug: Nab paclitaxel — Nab-Paclitaxel: 100mg/m2 on day 1, 8 and 15 every 4 weeks
  Other Names: Abraxane
  Arms: B: "Reduced dose (80%) combination-therapy strategy"

SUMMARY:
The aim of the study is to compare the efficacy and toxicity of full-dose Gemcitabine and reduced-dose combination chemotherapy in patients with non-resectable pancreatic cancer, who are unfit for full-dose combination chemotherapy.

The patients will be equally randomized to arm A or arm B:

Arm A: Full-dose single agent treatment with Gemcitabine 1000 mg/m2 weekly on days 1, 8,and 15 every 4 weeks.

Arm B: Reduced-dose (80%) combination-treatment with Gemcitabine plus Nab-Paclitaxel (Gemcitabine: 800 mg/m2 plus Nab-Paclitaxel: 100 mg/m2 on day 1, 8 and 15 every 4 weeks)

Progression-free survival, overall survival and response rate will be estimated for each group, as well as toxicity and quality of life will be prospectively registered.

DETAILED DESCRIPTION:
According to guidelines the recommended treatment for patients with non-resectable pancreatic cancer (PC) is combination chemotherapy, whereas old and/or fragile patients can be offered Gemcitabine monotherapy, if they are fit for treatment. Phase III trials show improved effect of combination chemotherapy compared to Gemcitabine, but these trials were restricted to fit patients younger than 75 years of age, as full-dose combination chemotherapy is more toxic.

Studies in colorectal cancer and a post-hoc analysis of Gemcitabine plus Nab-Paclitaxel in PC suggest that reduced-dose of combination chemotherapy may be more efficient in terms of progression-free survival and less toxic as compared to monotherapy in elderly and/or frail patients, but reduced start-dosing of GemNab is not currently labelled.

Moreover, a recent Danish register-based study showed that more use of combination chemotherapy at oncological departments was associated with improved outcome of patients with PC.

Elderly and frail patients with PC are in great need of better treatment results. Hence, a comparative study of reduced-dose combination chemotherapy is warranted and may be practice changing.

The aim of the study is to compare the efficacy and toxicity of full-dose Gemcitabine and reduced-dose combination chemotherapy in patients with non-resectable PC, who are unfit for full-dose combination chemotherapy.

The study is a national multicenter prospective randomized phase II trial, endorsed by the Danish Pancreas Cancer Group (DPCG). 98 patients with non-resectable PC, unfit for full-dose combination chemotherapy, but eligible for first-line chemotherapy, will be included.

The patients will be equally randomized to arm A or arm B:

Arm A: Full-dose single agent treatment with Gemcitabine 1000 mg/m2 weekly on days 1, 8 and 15 every 4 weeks.

Arm B: Reduced-dose (80%) combination-treatment with GemNab (Gemcitabine: 800 mg/m2 plus Nab-Paclitaxel: 100 mg/m2 on day 1, 8 and 15 every 4 weeks).

Progression-free survival, overall survival and response rate will be estimated for each group, as well as toxicity and quality of life will be prospectively registered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Adenocarcinoma of the pancreas, histopathologically or cytologically verified
* Non-resectable (locally advanced or metastatic) PC
* Patients unfit or not candidate for full-dose combination chemotherapy
* Patients eligible for full dose gemcitabine or reduced dose combination chemotherapy
* Performance status (PS) ≤2
* Measurable or non-measurable disease
* Adequate hematologic function defined as absolute neutrophil count (ANC) ≥1.5 x 10^9/l and platelets count ≥100x10^9/l within 2 weeks prior to enrollment
* Adequate organ function (bilirubin ≤1.5 x UNL (Upper Normal Limit) and eGFR (estimated Glomerular Filtration Rate) >50ml/min within 2 weeks prior to enrollment
* Toxicity of prior chemotherapy, including neurotoxicity, resolved to CTCAE <grade 2
* Oral and written informed consent must be obtained according to the local Ethics committee requirements
* Fertile patients must use adequate contraceptives

Exclusion Criteria:

* Patients eligible for downstaging/preoperative chemotherapy followed by resection or local ablation or irradiation
* Prior chemotherapy for PC (However, patients treated with adjuvant therapy with recurrence occurring more than 6 months after end of this treatment are eligible)
* Concurrent, non-curatively treated malignant neoplasm other than pancreatic adenocarcinoma
* Concurrent treatment with any other anti-cancer therapy
* Pregnant or breast-feeding patients
* Patients clearly intending to withdraw from the study if not randomized in the willing arm or patients who cannot be regularly followed up for psychological, social, familiar, or geographic reasons.
* Other condition or therapy, which in the investigator's opinion may pose a risk to the patient or interfere with the study objectives.
* Known allergy or intolerance to any of the drugs used in DPCG-01 (Gemcitabine, S1 or Nab-Paclitaxel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression Free Survival) | 1 year from end of study accrual.
  PFS is defined in the ITT population as the date of the randomization to the date of disease progression or date of death, whichever comes first. The date of PD is the date of scan, if progression is found on a CT scan, or date of visit at which clinical progression is found. PD at CT is defined according to RECIST version 1.1.

SECONDARY OUTCOMES:
OS (Overall Survival) | 1 year from end of study accrual.
  OS is defined in the ITT population as the date of randomization to date of death of all causes.
RR (Response rate) | 1 year from end of study accrual.
  In patients with measurable disease at baseline, RECIST version 1.1 will be used for evaluation of complete response (CR), partial response (PR), stable disease (SD) or PD. ORR will be calculated as the percentage of patients with CR+PR of all patients with measurable disease, who received at least one treatment and were evaluated by at least one diagnostic CT scan.
Hospitalizations | Through study completion, an average of 6 months.
  The total number of hospital admissions in a stationary unit with overnight stay from the start of treatment to the date of end of treatment will be assessed in the treated population. If the patient is readmitted for the same reason within 3 days (e.g., after weekend leave), this is not counted as a separate admission. The reasons for admission are registered as toxicity due to treatment or symptoms due to PC. The sum of hospitalizations is calculated for each randomization arm for comparison.
Quality of Life (QOL) assessed by EORTC QLQ-C30 at baseline and after 8, 16, and 24weeks | At baseline and at 8, 16, and 24 weeks.
  QoL scores collected will be linearly transformed to a scale of 0 to 100. Items will be grouped in health status scale (range 0 - 100, high is better), functional scales (range 0 - 100, high is better) and symptom scales (range 0 - 100, low is better). Each scale is summarized by its mean, and standard deviation for the patients in the two treatment groups. The difference in mean at 8, 16 and 24 weeks are compared with the baseline mean within in each treatment groups. The difference in mean between the treatment groups are compared at baseline, 8, 16 and 12 weeks.
Cumulative worst toxicity during treatment | From date of first treatment until 1 year from end of study treatment.
  (Adverse events ≥ grade 3 according to CTCAE version 5.0). All patients who have received 1 dose of chemotherapy will be calculated in the safety analyses. Cumulative worst toxicities ≥CTC grade 3 in the treated population are registered for each arm separately for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Ladekarl, Professor, Principal Investigator — Aalborg Universitets Hospital, Department of Oncology
Locations (1):
- Department of Oncology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen LS, Winther SB, Chen IM, Weber B, Ventzel L, Liposits G, Johansen JS, Detlefsen S, Egendal I, Shim S, Christensen S, Pfeiffer P, Ladekarl M. A randomized phase II study of full dose gemcitabine versus reduced dose gemcitabine and nab-paclitaxel in vulnerable patients with non-resectable pancreatic cancer (DPCG-01). BMC Cancer. 2023 Jun 16;23(1):552. doi: 10.1186/s12885-023-11035-6. PMID 37328835